CLINICAL TRIAL: NCT00525200
Title: p53-Adjusted Neoadjuvant Chemotherapy for Potentially Resectable Esophageal Cancer: A Multicenter, Randomized Controlled, Predictive Marker Clinical Trial
Brief Title: p53-Adjusted Neoadjuvant Chemotherapy for Potentially Resectable Esophageal Cancer
Acronym: PANCHO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daniela Kandioler (Other)
Collaborators: Medical University of Vienna (Other); Austrian Society Of Surgical Oncology (Other)
Responsible Party: Sponsor-Investigator, Daniela Kandioler, Univ. Prof. Dr., MBA, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ASSO OE-1; EudraCT 2006-006647-31
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Esophageal Cancer
Keywords: predictive marker; personalized therapy; response assessment; p53 genotype
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: 5-Fluoruracil, Cisplatinum
- B (Experimental)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: 5-Fluoruracil, Cisplatinum — 5 FU 1000mg/m2; days 1-5; 3 cycles: q21
  Cisplatin 80mg/m2; day 1; 3 cycles: q21
  Arms: A
Drug: Docetaxel — Docetaxel 75mg/m2, day 1; 3 cycles; q21
  Arms: B

SUMMARY:
Study Hypothesis:

PANCHO is a prospective randomized, predictive marker study, evaluating the interaction between the potential predictive marker 'p53 genotype' and response to induction chemotherapy in patients with esophageal cancer considered resectable.

170 patients with measurable disease will be enrolled in this study. After testing the marker genotype (two genotypes: p53 normal or p53 mutant) patients will be stratified according to histological subtype only (adeno- or squamous cell carcinoma) and will be randomly assigned to receive 3 cycles of either 5-fluorouracil (5FU)/cisplatin or docetaxel monotherapy as neoadjuvant therapy. All patients will be rendered to subsequent surgery in order to assess both clinical and pathohistological response.

DETAILED DESCRIPTION:
PANCHO will test the hypothesis that p53 genotype is predictive for response to chemotherapy. The study uses the marker by treatment interaction design. In this design, we assume that the status of the marker splits the whole population into two distinct groups (p53 normal versus p53 mutant).

Patients in each marker group are randomly assigned to two different treatments, and planned statistical analysis is to test whether one treatment is superior to the other within each marker group separately.

The marker information but not the treatment is blinded to the patient and the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Histological verification of esophageal cancer
* Presence of T2,T3,T4 or any N1 (except M1)
* Clinically measurable lesions according to RECIST criteria
* Males and females, age >18 to 75 or older with WHO performance status 1
* No prior tumor therapy for esophageal cancer
* No other malignancy in history within 5 years before evaluation
* Performance status of 0-2 on ECOG scale
* Medical fitness (adequate for possible esophageal resection, adequate organ function: see protocol)
* Signed informed consent
* Males and females with reproductive potential must use an approved contraceptive method. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Inoperability (technical or functional)
* Clinical stage cT1N0, any M1
* Treatment with any of the investigational drugs within the last 6 months
* Concurrent administration of any other tumor therapy
* Pregnancy, breast feeding
* Serious concomitant disorders that would compromise the safety of the patient or ability to complete the study
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tumor response (clinical and pathological) to neoadjuvant treatment in relation to p53 genotype | 12 weeks

SECONDARY OUTCOMES:
Complete pathological response and relation to p53 genotype | 12 weeks
Complete tumor resection rate | 12 weeks
Perioperative morbidity and mortality | 16 weeks
Disease free and overall survival and relation to p53 genotype | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Kandioler, Prof., MBA, Study Chair — ASSO Representative, MUW, p53research Head; Johannes Zacherl, Prof., Study Director — Medical University of Vienna, MUV; Michael Hejna, Prof., Study Director — MUW
Locations (13):
- Austria (13):
  - Landesklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Landesklinikum Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Rudolfstiftung, Vienna, Vienna
  - SMZ OST, Vienna, Vienna
  - Wilhelminenspital, Vienna, Vienna
  - Landesklinikum Feldkirch, Feldkirch, Vorarlberg
  - Landeskrankenhaus Leoben, Leoben
  - Krankenhaus der Elisabethinen, Linz
  - Krankenhaus der Barmherzigen Brüder, Stankt Veit
  - Medical University of Vienna, Vienna
  - Kaiser Franz Josef Spital, Vienna
  - Hanusch Krankenhaus, Vienna

REFERENCES:
- [Background] Kandioler D et al. p53 adapted neoadjuvant therapy for esophageal cancer: pilot study. JCO, vol 25, 18S: 206s
- See also: p53research group at the University of Vienna — http://www.p53.at